CLINICAL TRIAL: NCT01171495
Title: Phase 3 Study That Assesses the Impact of a Nutrition Intervention on HIV/AIDS Infected Patients: Kingston, Jamaica
Brief Title: Impact of Nutrition Intervention on HIV/AIDS Infected Patients
Acronym: INI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Caribbean Health Research Council (Other)
Collaborators: The University of The West Indies (Other)
Responsible Party: Sharon Dawson, Ministry of Health,Kingston, Jamaica and The University of the West Indies, Mona, Jamaica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHRC 51016
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-02

CONDITIONS: Human Immunodeficiency Virus (HIV); Acquired Immune Deficiency Syndrome (AIDS)
Keywords: HIV/AIDS; Nutrition Therapy; Dietary Supplement; Antioxidant; Immunity; CD4 count; Anthropometry; Body Mass Index
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Theragran-M

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ensure Plus + Multivitamin/Counselling (Experimental)
  Interventions: Dietary Supplement: Theragran-M; Ensure Plus
- Multivitamin/Counselling (Active Comparator)
  Interventions: Dietary Supplement: Theragran-M

INTERVENTIONS:
Dietary Supplement: Theragran-M; Ensure Plus — Theragran-M: One tablet daily for 6-months. Ensure Plus: One 8 fl.oz. bottle daily for 6-months. Nutritional counselling: at baseline, and at monthly follow-up visits.
  Arms: Ensure Plus + Multivitamin/Counselling
Dietary Supplement: Theragran-M — Theragran-M: One tablet daily for 6-months. Nutritional counselling: at baseline and at monthly follow-up visits.
  Arms: Multivitamin/Counselling

SUMMARY:
Intervention to investigate the efficacy of a nutritional supplement among ARV-naïve, asymptomatic HIV positive patients with a CD4 count in the range 300-550 cells/ul.

DETAILED DESCRIPTION:
To investigate the efficacy of a nutritional supplement among ARV-naïve, asymptomatic HIV positive patients with a CD4 count in the range 300-550 cells/ul.

A total of 120 participants will be stratified by age and gender and randomly assigned to two treatment arms. Sixty (60) participants will be assigned to receive dietary counselling and a multivitamin/mineral supplement, with sixty (60) additionally receiving an oral Medical Nutritional Supplement (MNS).

Participants will be followed for six months post-randomization: at baseline, 3 months and 6 months. The principal outcome measure is Body Mass Index, used as a proxy for 'nutritional status'. Secondary outcome measures include immune status and antioxidant status.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive individuals in the age range 18 to 50 years.
* Individuals whose CD4 count was between 300-550 cells/uL.
* Individuals who met the study criteria and were interested in being enrolled.
* Individuals not on ARV therapy.
* Women who were not pregnant.

Exclusion Criteria:

* On the clinician's advice, individuals could be excluded from enrollment.
* Individuals who were unable to carry out the study intervention e.g. homeless, impaired mental state etc.
* Individuals who were unlikely to complete follow-up based on pre-enrolment assessment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2008-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Effects of nutritional intervention on anthropometry in HIV infected individuals. | 6 months
  Body Mass Index

SECONDARY OUTCOMES:
Effects of nutritional intervention on the clinical and immune status in HIV infected individuals. | 6 months
  Immune status (CD4 cell count, total lymphocyte count), antioxidant status.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon M Dawson, MSc, Principal Investigator — University of the West Indies, Mona ,Jamaica, West Indies
Locations (1):
- Comprehensive Health Centre, Kingston, Jamaica